CLINICAL TRIAL: NCT05922410
Title: Different Maxillary Sinus 3D Shapes Assessment Using CBCT Volumetric Segmentation: A Cross Sectional Study
Brief Title: Different Maxillary Sinus 3D Shapes Assessment Using CBCT Volumetric Segmentation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Jasmine Mohammed Aly, SPECIALIST PHD candidate, Cairo University
Other Study IDs: ORAD 7 - 1 - 1
Record Dates: First submitted 2023-06-08; First posted 2023-06-28 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Cone-beam Computed Tomography; Maxillary Sinus; Anatomical Variations

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: cone beam computed tomography — cone beam computed tomography
  Other Names: CBCT

SUMMARY:
the study aims to assist the different 3D shapes of maxillary sinus in adult individuals among Egyptian population,The data collection will be obtained from the data base available at the department of Oral and Maxillofacial Radiology, Faculty of Dentistry, Cairo University. CBCT images will be obtained from Egyptian patients who were referred to the CBCT unit in oral and maxillofacial radiology department for different purposes. The following radiographic examination will be done in Oral and Maxillofacial Radiology Department, Faculty Dentistry, Cairo University. semiautomated segmentation will be performed for the maxillary sinus in both side and then linear and 3D volume will be assessed for each sinus.

ELIGIBILITY:
Inclusion Criteria:

* CBCT scans of adult Egyptian patients, males and females, with age range between 18 and 50 years old. Patients will be divided into two age groups (group 1 less than or equal 30 years old, group2 more than 30 years old).
* CBCT scans of patient without previous orthodontic treatment.
* CBCT scans without any other treatment that might interfere with the natural course of maxillomandibular growth and development.

Exclusion Criteria:

-Scans with maxillary pathologies like (tumors, odontogenic lesions, bone lesions).

* Patients with traumatic injuries or fractures affecting the maxillary sinus.
* Patients with missing upper premolar or molar teeth in one side or both sides.
* Patients with skeletal asymmetries, craniofacial traumas and developmental anomalies such as palatal cleft.
* Images of low-resolution quality.
* Distortion of images or presence of any artifacts.

Ages: 20 Years to 50 Years | Sex: All
Age Groups: Adult
Study Population: CBCT maxillofacial scans belonging to Egyptian individuals will be examined
Sampling Method: Probability Sample
Enrollment: 29 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2023-08-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of different volumetric 3D shapes of maxillary sinus | 1 year
  Assessment of different volumetric 3D shapes of maxillary sinus

SECONDARY OUTCOMES:
Symmetrical assessment of maxillary sinus volumetric 3D shape in both sides in the same individual | 1 year
  Symmetrical assessment of maxillary sinus volumetric 3D shape in both sides in the same individual
Maxillary sinus volumetric 3D Shape with sex variables | 1 year
  Maxillary sinus volumetric 3D Shape with sex variables